CLINICAL TRIAL: NCT00848029
Title: Safety and Immunogenicity of Two Doses of Monovalent Inactivated Influenza Vaccine That is Adjuvanted With MF59C.1 (MF59) and Uses a Surface Antigen From a Potential Pandemic Virus Strain Candidate (H5N1) in Adult and Elderly Subjects Using Four Different Vaccination Schedules
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V87P12; 2008-003008-72
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2011-12

CONDITIONS: Pre-pandemic Influenza Vaccine
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Monovalent inactivated influenza vaccine

INTERVENTIONS:
Biological: Monovalent inactivated influenza vaccine — Two doses of monovalent inactivated influenza adjuvanted vaccine

SUMMARY:
The present study will evaluate the immunogenicity, safety and immunogenicity of two doses of monovalent inactivated influenza vaccine that is adjuvanted with MF59C.1 (MF59) and uses a surface antigen from a potential pandemic virus strain candidate (H5N1) in Adult Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 to 60 years of age who are mentally competent and who have signed an informed consent form after having received a detailed explanation of the study protocol;
* In good health as determined by:

  * Medical history,
  * Physical examination,
  * Clinical judgment of the Investigator;
* Able to understand and comply with all study procedures and to complete study diaries, can be contacted, and will be available for all study visits.

Exclusion Criteria:

* Previous receipt of any H5 vaccine;
* Receipt of another investigational agent within 4 weeks, or before completion of the safety follow-up period in another study, whichever is longer, prior to enrollment and unwilling to refuse participation in another clinical study through the end of the study;
* Experienced any acute disease or infection requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis is acceptable) within the past 7 days;
* Experienced fever (defined as axillary temperature 38.0°C) within 3 days prior to Visit 1;
* Pregnant or breastfeeding;
* Females of childbearing potential who refuse to use an acceptable method of birth control for the duration of the study. Adequate contraception is defined as hormonal (e.g., oral, injection, transdermal patch, implant, cervical ring), barrier (e.g., condom with spermicide or diaphragm with spermicide), intrauterine device (e.g., IUD), or monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject's study entry;
* Any serious disease, such as:

  * cancer,
  * Autoimmune disease,
  * diabetes mellitus,
  * chronic pulmonary disease,
  * acute or progressive hepatic disease,
  * acute or progressive renal disease;
* Surgery planned during the study period;
* Bleeding diathesis;
* Hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the study vaccine;
* History of any neurological symptoms or signs following administration of any vaccine, or anaphylactic shock following administration of any vaccine;
* Known or suspected impairment/alteration of immune function, for example, resulting from:

  * Receipt of immunosuppressive therapy (any corticosteroid therapy
  * Receipt of immunostimulants,
  * High risk for developing an immunocompromising disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of antibody response to a monovalent inactivated influenza vaccine adjuvanted with MF59 and uses a surface antigen from a potential pandemic homologous virus strain candidate (H5N1). | 6 months

SECONDARY OUTCOMES:
Evaluation of safety of the monovalent inactivated influenza vaccine that is adjuvanted with MF59C.1 (MF59) and uses a surface antigen from a potential pandemic virus strain candidate (H5N1) in Adult Subjects. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Vaccination and Travel Medicine Centre, Hradec Králové, Czechia

REFERENCES:
- [Result] Beran J, Abdel-Messih IA, Raupachova J, Hobzova L, Fragapane E. A phase III, randomized, open-label study to assess the tolerability and immunogenicity of an H5N1 influenza vaccine administered to healthy adults with a 1-, 2-, 3-, or 6-week interval between first and second doses. Clin Ther. 2010 Dec;32(13):2186-97. doi: 10.1016/S0149-2918(11)00024-5. PMID 21316535